CLINICAL TRIAL: NCT04472286
Title: Healthy Bones, Healthy Life: Effect of Habitual Physical Activity on Bone and Metabolic Health in Pediatric Cancer Survivors
Brief Title: Healthy Bones, Healthy Life: Habitual Physical Activity on Bone & Metabolic Health in Pediatric Cancer Survivors
Acronym: HBHL
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0206-20-FB
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric; Pediatric ALL; Pediatric Lymphoma; Bone Loss; Metabolic Syndrome; Habitual Physical Activity; Precursor Cell Lymphoblastic Leukemia; Lymphoma; Leukemia; Lymphoid Leukemia; Pediatric; Osteoporosis; Osteoporosis Risk
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Bone Diseases, Metabolic; Metabolic Syndrome; Lymphoma; Leukemia; Leukemia, Lymphoid; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Cancer Survivors: Children and adolescents who have completed treatment of for acute lymphoblastic leukemia (ALL) and lymphoma.

SUMMARY:
This project will examine habitual physical activity, bone health, and insulin resistance in pediatric acute lymphocytic leukemia (ALL) and lymphoma cancer survivors at two time points: baseline and 6 months. At the two study timepoints, all study participants will be asked to wear an accelerometer, receive a DXA scan of the lumbar spine and hip, and have blood drawn for analysis. Study participants will be given a gift card stipend for each study visit attended. Study visits will coincide with regular office visits to Children's Hospital Oncology Clinic and the Children's Hospital Survivorship Clinics whenever possible. The potential mechanism by which physical activity mediates bone changes will be explored by concurrently measuring changes in lean/fat mass and metabolic status. This pilot study will provide data to inform the design of a randomized controlled trial to test the effect of a physical activity intervention on bone health in PCS.

DETAILED DESCRIPTION:
Childhood cancer treatments are increasingly effective, leading to dramatic improvements in survival rates. These treatments often have devastating effects on the overall health of pediatric cancer survivors (PCS) since they occur during a critical time of bone growth, including increased risks of poor bone health, fracture, and diabetes. In normal child development, physical activity habits influence bone density and structure, which affect bone strength in adulthood. Despite this well-understood principle of bone development, there are no exercise guidelines for improving bone health in PCS. The long-term goal of this research is to develop an effective exercise intervention to improve bone health after cancer therapy. As a first step, the investigators propose to test the hypothesis that the intensity and amount of ground impact of a child's daily physical activity will influence changes in bone density in PCS. The Specific Aims are to (1) examine the effect of physical activity on lumbar bone density of PCS and to (2) evaluate how physical activity influences bone density. In a prospective cohort study, the investigators will enroll 38 pediatric and adolescent survivors (ages 5-18) of acute lymphoblastic leukemia or lymphoma at any post-treatment time point. Aim 1: At two assessments, baseline and six months later, bone density and structure (by DXA scan, a type of x-ray that can measure bone density and the amount of muscle and fat in the body) and physical activity level (by accelerometry, a device like a fitness tracker) will be evaluated. Each child will be categorized as having low or high physical activity based on accelerometry measures averaged from baseline and six-month assessments. Bone changes (0-6 months) will be compared between low and high activity groups. Aim 2: Evaluate potential mechanisms by which physical activity mediates changes in bone, including the effects of lean mass (measured by DXA) and metabolic health (lipid panel, insulin sensitivity (HOMA-IR, hemoglobin A1c), vitamin D). Long-term impact: This research will provide information as to the types of exercise that impact bone health in PCS. This study will help develop effective, evidence-based exercise therapies. These therapies may help prevent fractures and associated disability, leading to an improvement in the quality of life for survivors of pediatric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 5-18
2. Diagnosis of ALL or Lymphoma
3. Between 1-13 months post-cancer treatment

Exclusion Criteria:

1. Children younger than 5 years old or 19 or older
2. Children without a diagnosis of ALL or lymphoma
3. Children receiving ongoing cancer treatment
4. Children with Down syndrome (identified as a precancerous condition affecting BMD)
5. Children with a prior history of bisphosphonate use or other medication directed at increasing bone density

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric cancer survivors who are in the first year after treatment completion
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (g/cm2) | 6 months
  z-score of lumbar Spine bone density- DXA scan
Hip structural analysis | 6 months
  DXA scan
Physical Activity Level | 6 months
  Physical Activity as measured by accelerometry

SECONDARY OUTCOMES:
Lipid panel | 6 months
  cholesterol (total, HDL, and LDL) and triglycerides will be measured, which are an indicator of overall cardiovascular health which can impact insulin sensitivity
Homeostatic Model Assessment for Insulin Resistance | 6 months
  Fasting Insulin and Fasting Glucose will be combined to calculate the HOMA-IR, which is an indicator of insulin sensitivity
Hemoglobin A1c | 6 months
  measure of the glycated hemoglobin in blood, which is an indicator of insulin sensitivity
Vitamin D | 6 months
  measures the levels of vitamin D in the blood which is an indicator of bone health

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Bilek, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No